CLINICAL TRIAL: NCT05578118
Title: Physical, Mental, and Motor Development of Children Born From Intracytoplasmic Sperm Injection With Assisted Oocyte Activation With Calcium Ionophore
Brief Title: Health of Children Born From ICSI With AOA (AOA-BABIES)
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10/22/DD-BVMD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2023-08

CONDITIONS: Infertility; Intracytoplasmic Sperm Injection
Keywords: ICSI; Total fertilization failure; AOA; ASQ-3; Health of children
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICSI + AOA: Children born after ICSI + AOA
- Control: Children born after ICSI

SUMMARY:
The investigators follow up on the development of children born from ICSI-AOA using the Developmental Red Flags and Ages & Stages Third Edition (ASQ-3) Questionnaires to give strong evidence about the safety of AOA in assisted reproductive technology.

DETAILED DESCRIPTION:
Intracytoplasmic sperm injection (ICSI) is the most widely utilized assisted reproductive technique (ART) worldwide. Fertilization rates obtained after ICSI treatment are reported between 70 and 80%, representing the most efficient ART; however, complete post-ICSI fertilization failure still occurs in 3-5% of cases.

The leading cause of failed fertilization is failure to achieve oocyte activation, a crucial stage in the initiation of embryo development during fertilization. Assisted oocyte activation (AOA) using a calcium ionophore has been used for over a decade following ICSI fertilization failure. AOA is not considered a routine practice of ART yet, which is only suitable for patients with proper indications, including (i) total fertilization failure or low fertilization rate (<30%) in the previous IVF; (ii) severe male factor infertility; (iii) patients with a history of embryo arrest or poor embryo quality in previous IVF cycle.

Regarding technique, the artificial rise of induced calcium rises cannot precisely mimic the physiologically sperm-induced calcium oscillations. Little is known yet about the possible adverse effects of ionophores on post-implantation embryo development. Numerous studies have been conducted to compare the development of children born from ICSI - AOA versus non-AOA. Thus, the investigators performed this study to investigate the physical, mental, and motor development of children born following ICSI - AOA using the Developmental Red Flags and Ages & Stages Third Edition (ASQ-3) Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

All single, live babies born following ICSI with AOA and ICSI without AOA from 08/2020 to 04/2021.

Parents consent to participate in the study. Group ICSI+AOA: Embryos from ICSI with AOA with calcium ionophore

In the ICSI+AOA group, indications of AOA are:

* Previous failed IVF treatment with no fertilization or poor fertilization rate (fertilized oocytes/pick-up oocytes<35%) or poor embryo result (number of embryos/pick-up oocytes<35%, <3 embryos, no good-quality embryo)
* Using sperm after retrieval technique, cryptozoospermia Group Control: Embryos from ICSI without AOA.

In the Control group, the indications of AOA for the next IVF cycle (if patients continue the next IVF cycle) are:

* Currently failed IVF treatment with no fertilization or poor fertilization rate (fertilized oocytes/pick-up oocytes<35%) or poor embryo result (number of embryos/pick-up oocytes<35%, <3 embryos, no good-quality embryo)

Exclusion Criteria:

Embryos with PGT. Oocyte donation

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In the ICSI+AOA group, indications of AOA are:
  * Previous failed IVF treatment with no fertilization or poor fertilization rate (fertilized oocytes/pick-up oocytes<35%) or poor embryo result (number of embryos/pick-up oocytes<35%, <3 embryos, no good-quality embryo)
  * Using sperm after retrieval technique, cryptozoospermia
  In the Control group, the indications of AOA for the next IVF cycle (if patients continue the next IVF cycle) are:
  * Currently failed IVF treatment with no fertilization or poor fertilization rate (fertilized oocytes/pick-up oocytes<35%) or poor embryo result (number of embryos/pick-up oocytes<35%, <3 embryos, no good-quality embryo)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The percentage of abnormal ASQ-3 score | 12 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross Motor, Fine Motor, Problem-solving, and Personal-Social Each element has 6 questions. If the answer is Yes, score = 10, Sometimes = 5, and Not yet = 0.
  ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | 12 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Gross motor | 12 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Fine motor | 12 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Problem-solving skill | 12 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Personal-Social | 12 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
The rate of children who have at least one red flag sign(s): | 12 months after birth
  For children at 12 months: they
  * No response when being called by their name
  * Does not understand "no"
  * Can not stand even when being supported
  * Apathy or non-observance of the caregiver
  * Does not look at the point where the caregiver points
Duration of breastfeeding | 12 months after birth
  Duration of breastfeeding
Infant age at which weaning starts | 12 months after birth
  Infant age at which weaning starts
Name of diseases that lead to hospital admission | 12 months after birth
  Name of diseases that lead to hospital admission
Number of hospital admission | 12 months after birth
  Number of hospital admission
Weight | 12 months after birth
  Weight on the examination date
Height | 12 months after birth
  Height on the examination date

OTHER OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery
Mode of delivery | At birth
  Vaginal birth or C-section
Birth weight | At birth
  Weight of baby born
Length circumference | At birth
  Length circumference after birth
Head circumference | At birth
  Head circumference after birth
Rate of congenital anomalies | At birth
  Any congenital anomalies detected in baby born
Length of neonatal intensive care unit (NICU) admission | Up to 28 days after birth
  Number of admission days to NICU
Rate of Respiratory distress syndrome | Up to 28 days after birth
  Respiratory distress syndrome (RDS), diagnosed as the presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Rate of Periventricular haemorrhage | Up to 28 days after birth
  Periventricular haemorrhage II B or worse, will be diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al.
Rate of Necrotizing enterocolitis | Up to 28 days after birth
  Necrotizing enterocolitis (NEC) will be diagnosed according to Bell.
Rate of Proven sepsis | Up to 28 days after birth
  Proven sepsis, will be diagnosed on the combination of clinical signs and positive blood cultures.
Rate of Composite of poor perinatal outcomes | Up to 28 days after birth
  Composite of poor perinatal outcomes, defined as intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis.
Rate of long-term illness and chronic conditions | Up to 28 days after birth
  Any long-term illness and chronic condition appears in a child.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Vuong Ngoc, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alberio R, Zakhartchenko V, Motlik J, Wolf E. Mammalian oocyte activation: lessons from the sperm and implications for nuclear transfer. Int J Dev Biol. 2001 Oct;45(7):797-809. PMID 11732839
- [Result] Bos-Mikich A, Whittingham DG, Jones KT. Meiotic and mitotic Ca2+ oscillations affect cell composition in resulting blastocysts. Dev Biol. 1997 Feb 1;182(1):172-9. doi: 10.1006/dbio.1996.8468. PMID 9073459
- [Result] Capalbo A, Ottolini CS, Griffin DK, Ubaldi FM, Handyside AH, Rienzi L. Artificial oocyte activation with calcium ionophore does not cause a widespread increase in chromosome segregation errors in the second meiotic division of the oocyte. Fertil Steril. 2016 Mar;105(3):807-814.e2. doi: 10.1016/j.fertnstert.2015.11.017. Epub 2015 Dec 1. PMID 26658129
- [Result] D'haeseleer E, Vanden Meerschaut F, Bettens K, Luyten A, Gysels H, Thienpont Y, De Witte G, Heindryckx B, Oostra A, Roeyers H, Sutter PD, van Lierde K. Language development of children born following intracytoplasmic sperm injection (ICSI) combined with assisted oocyte activation (AOA). Int J Lang Commun Disord. 2014 Nov;49(6):702-9. doi: 10.1111/1460-6984.12100. Epub 2014 May 26. PMID 24861451
- [Result] Ducibella T, Huneau D, Angelichio E, Xu Z, Schultz RM, Kopf GS, Fissore R, Madoux S, Ozil JP. Egg-to-embryo transition is driven by differential responses to Ca(2+) oscillation number. Dev Biol. 2002 Oct 15;250(2):280-91. PMID 12376103
- [Result] Ebner T, Oppelt P, Wober M, Staples P, Mayer RB, Sonnleitner U, Bulfon-Vogl S, Gruber I, Haid AE, Shebl O. Treatment with Ca2+ ionophore improves embryo development and outcome in cases with previous developmental problems: a prospective multicenter study. Hum Reprod. 2015 Jan;30(1):97-102. doi: 10.1093/humrep/deu285. Epub 2014 Nov 5. PMID 25376461
- [Result] Fawzy M, Emad M, Mahran A, Sabry M, Fetih AN, Abdelghafar H, Rasheed S. Artificial oocyte activation with SrCl2 or calcimycin after ICSI improves clinical and embryological outcomes compared with ICSI alone: results of a randomized clinical trial. Hum Reprod. 2018 Sep 1;33(9):1636-1644. doi: 10.1093/humrep/dey258. PMID 30099496
- [Result] Heytens E, Soleimani R, Lierman S, De Meester S, Gerris J, Dhont M, Van der Elst J, De Sutter P. Effect of ionomycin on oocyte activation and embryo development in mouse. Reprod Biomed Online. 2008 Dec;17(6):764-71. doi: 10.1016/s1472-6483(10)60403-8. PMID 19079959
- [Result] Hirata, K., Nakamura, Y., Hattori, H., Kuchiki, M., Sakamoto, E., & Kyono, K. (2013). Follow-up child growth regarding new technologies: Testicular sperm extraction (TESE), in vitro maturation (IVM), and assisted oocyte activation (AOA). Fertility and Sterility, 100(3), S470. https://doi.org/10.1016/j.fertnstert.2013.07.445
- [Result] Kashir J, Nomikos M, Lai FA, Swann K. Sperm-induced Ca2+ release during egg activation in mammals. Biochem Biophys Res Commun. 2014 Aug 1;450(3):1204-11. doi: 10.1016/j.bbrc.2014.04.078. Epub 2014 Apr 21. PMID 24769204
- [Result] Kim BY, Yoon SY, Cha SK, Kwak KH, Fissore RA, Parys JB, Yoon TK, Lee DR. Alterations in calcium oscillatory activity in vitrified mouse eggs impact on egg quality and subsequent embryonic development. Pflugers Arch. 2011 May;461(5):515-26. doi: 10.1007/s00424-011-0955-0. Epub 2011 Mar 23. PMID 21431324
- [Result] Koo OJ, Jang G, Kwon DK, Kang JT, Kwon OS, Park HJ, Kang SK, Lee BC. Electrical activation induces reactive oxygen species in porcine embryos. Theriogenology. 2008 Oct 15;70(7):1111-8. doi: 10.1016/j.theriogenology.2008.06.031. PMID 18675447
- [Result] Miller N, Biron-Shental T, Sukenik-Halevy R, Klement AH, Sharony R, Berkovitz A. Oocyte activation by calcium ionophore and congenital birth defects: a retrospective cohort study. Fertil Steril. 2016 Sep 1;106(3):590-596.e2. doi: 10.1016/j.fertnstert.2016.04.025. Epub 2016 Apr 30. PMID 27143515
- [Result] Ozil JP, Huneau D. Activation of rabbit oocytes: the impact of the Ca2+ signal regime on development. Development. 2001 Mar;128(6):917-28. doi: 10.1242/dev.128.6.917. PMID 11222146
- [Result] Ozil JP, Banrezes B, Toth S, Pan H, Schultz RM. Ca2+ oscillatory pattern in fertilized mouse eggs affects gene expression and development to term. Dev Biol. 2006 Dec 15;300(2):534-44. doi: 10.1016/j.ydbio.2006.08.041. Epub 2006 Aug 25. PMID 16996050
- [Result] Swann K, Ozil JP. Dynamics of the calcium signal that triggers mammalian egg activation. Int Rev Cytol. 1994;152:183-222. doi: 10.1016/s0074-7696(08)62557-7. No abstract available. PMID 8206704
- [Result] Eftekhar M, Janati S, Rahsepar M, Aflatoonian A. Effect of oocyte activation with calcium ionophore on ICSI outcomes in teratospermia: A randomized clinical trial. Iran J Reprod Med. 2013 Nov;11(11):875-82. PMID 24639711
- [Result] Tesarik J, Sousa M. Key elements of a highly efficient intracytoplasmic sperm injection technique: Ca2+ fluxes and oocyte cytoplasmic dislocation. Fertil Steril. 1995 Oct;64(4):770-6. doi: 10.1016/s0015-0282(16)57853-4. PMID 7672149
- [Result] Vanden Meerschaut F, Leybaert L, Nikiforaki D, Qian C, Heindryckx B, De Sutter P. Diagnostic and prognostic value of calcium oscillatory pattern analysis for patients with ICSI fertilization failure. Hum Reprod. 2013 Jan;28(1):87-98. doi: 10.1093/humrep/des368. Epub 2012 Oct 18. PMID 23081875
- [Result] Vanden Meerschaut F, Nikiforaki D, De Roo C, Lierman S, Qian C, Schmitt-John T, De Sutter P, Heindryckx B. Comparison of pre- and post-implantation development following the application of three artificial activating stimuli in a mouse model with round-headed sperm cells deficient for oocyte activation. Hum Reprod. 2013 May;28(5):1190-8. doi: 10.1093/humrep/det038. Epub 2013 Mar 12. PMID 23482335
- [Result] Vanden Meerschaut F, Nikiforaki D, Heindryckx B, De Sutter P. Assisted oocyte activation following ICSI fertilization failure. Reprod Biomed Online. 2014 May;28(5):560-71. doi: 10.1016/j.rbmo.2014.01.008. Epub 2014 Jan 31. PMID 24656559
- [Result] WHO child growth standards: Length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age: Methods and development. (n.d.). Retrieved June 10, 2022, from https://www.who.int/publications-detail-redirect/924154693X
- [Result] Yoshida S, Plant S. Mechanism of release of Ca2+ from intracellular stores in response to ionomycin in oocytes of the frog Xenopus laevis. J Physiol. 1992 Dec;458:307-18. doi: 10.1113/jphysiol.1992.sp019419. PMID 1302268